CLINICAL TRIAL: NCT07043452
Title: Measuring Acute Drug Demand in Humans II
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The lead investigator moved institutions and the study will not continue upon his departure.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00454735
Record Dates: First submitted 2025-06-09; First posted 2025-06-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Central Nervous System Stimulants; Cannabinoids; Benzodiazepines; Analgesics, Opioid; Nonprescription Drugs; Dosage Forms

STUDY DESIGN:
Intervention Model Description: This study will use a fully within subjects design (i.e., all subjects were to receive all drug combination conditions in a latin-square randomized order).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Experimental Session 1 (Experimental): This is the single arm that will go through all within-subject dose conditions in a Latin-Square randomized order.
  Interventions: Drug: Blinded Study Medication - Condition 1
- Experimental Session 2 (Experimental): This is the single arm that will go through all within-subject dose conditions in a Latin-Square randomized order.
  Interventions: Drug: Blinded Study Medication - Condition 2
- Experimental Session 3 (Experimental): This is the single arm that will go through all within-subject dose conditions in a Latin-Square randomized order.
  Interventions: Drug: Blinded Study Medication - Condition 3
- Experimental Session 4 (Experimental): This is the single arm that will go through all within-subject dose conditions in a Latin-Square randomized order.
  Interventions: Drug: Blinded Study Medication - Condition 4
- Experimental Session 5 (Experimental): This is the single arm that will go through all within-subject dose conditions in a Latin-Square randomized order.
  Interventions: Drug: Blinded Study Medication - Condition 5
- Experimental Session 6 (Experimental): This is the single arm that will go through all within-subject dose conditions in a Latin-Square randomized order.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Blinded Study Medication - Condition 1 — Participants will receive a double-blinded oral study medication as part of the participant's experimental sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, the medications are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study). Participants may receive a study drug that contains a prescription stimulant, a prescription cannabinoid (related to the active ingredient in cannabis or marijuana), a benzodiazepine (e.g., anti- anxiety medication), an opioid (e.g., a pain medication), a sleep medication, and/or an over-the-counter medication. The study is deeply blinded so that participants are not aware of possible drug conditions in the study and indication of the study drug names in the clinicaltrials.gov record would comprise the blind of the study. Detailed drug condition information will be added upon completion of study.
  Other Names: stimulant; cannabinoid; benzodiazepine; opioid; sleep medication; over the counter (OTC) medication
  Arms: Experimental Session 1
Drug: Blinded Study Medication - Condition 2 — Participants will receive a double-blinded oral study medication as part of the participant's experimental sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, the medications are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study). Participants may receive a study drug that contains a prescription stimulant, a prescription cannabinoid (related to the active ingredient in cannabis or marijuana), a benzodiazepine (e.g., anti- anxiety medication), an opioid (e.g., a pain medication), a sleep medication, and/or an over-the-counter medication. The study is deeply blinded so that participants are not aware of possible drug conditions in the study and indication of the study drug names in the clinicaltrials.gov record would comprise the blind of the study. Detailed drug condition information will be added upon completion of study.
  Other Names: stimulant; cannabinoid; benzodiazepine; opioid; sleep medication; over-the-counter (OTC) medication
  Arms: Experimental Session 2
Drug: Blinded Study Medication - Condition 3 — Participants will receive a double-blinded oral study medication as part of the participant's experimental sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, the medications are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study). Participants may receive a study drug that contains a prescription stimulant, a prescription cannabinoid (related to the active ingredient in cannabis or marijuana), a benzodiazepine (e.g., anti- anxiety medication), an opioid (e.g., a pain medication), a sleep medication, and/or an over-the-counter medication. The study is deeply blinded so that participants are not aware of possible drug conditions in the study and indication of the study drug names in the clinicaltrials.gov record would comprise the blind of the study. Detailed drug condition information will be added upon completion of study.
  Other Names: stimulant; cannabinoid; benzodiazepine; opioid; sleep medication; over-the-counter (OTC) medication
  Arms: Experimental Session 3
Drug: Blinded Study Medication - Condition 4 — Participants will receive a double-blinded oral study medication as part of the participant's experimental sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, the medications are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study). Participants may receive a study drug that contains a prescription stimulant, a prescription cannabinoid (related to the active ingredient in cannabis or marijuana), a benzodiazepine (e.g., anti- anxiety medication), an opioid (e.g., a pain medication), a sleep medication, and/or an over-the-counter medication. The study is deeply blinded so that participants are not aware of possible drug conditions in the study and indication of the study drug names in the clinicaltrials.gov record would comprise the blind of the study. Detailed drug condition information will be added upon completion of study.
  Other Names: stimulant; cannabinoid; benzodiazepine; opioid; sleep medication; over-the-counter (OTC) medication
  Arms: Experimental Session 4
Drug: Blinded Study Medication - Condition 5 — Participants will receive a double-blinded oral study medication as part of the participant's experimental sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, the medications are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study). Participants may receive a study drug that contains a prescription stimulant, a prescription cannabinoid (related to the active ingredient in cannabis or marijuana), a benzodiazepine (e.g., anti- anxiety medication), an opioid (e.g., a pain medication), a sleep medication, and/or an over-the-counter medication. The study is deeply blinded so that participants are not aware of possible drug conditions in the study and indication of the study drug names in the clinicaltrials.gov record would comprise the blind of the study. Detailed drug condition information will be added upon completion of study.
  Other Names: stimulant; cannabinoid; benzodiazepine; opioid; sleep medication; over-the-counter (OTC) medication
  Arms: Experimental Session 5
Drug: Placebo — Double blind administration of placebo.
  Arms: Experimental Session 6

SUMMARY:
This research is being done to evaluate the impact of various drugs and combinations of drugs on mood, pain, and performance.

DETAILED DESCRIPTION:
This research is being done to evaluate the impact of various drugs and combinations of drugs on mood, pain, and performance. Participants will complete 1 screening visit and 7 study test sessions. During the study sessions the participant will receive a study drug that may contain blinded drugs or drug combinations. Participants will answer questions about how the participant feels, perform tasks that measure the participant's cognitive ability and experience of pain, and have heart rate and blood pressure measured. While not at the laboratory, participants will be asked to wear a wristwatch that measures sleep and activity and complete questions about sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-55 years
2. Vital signs in normal range as reviewed by study medical team
3. Person is willing and able to provide informed consent

Exclusion Criteria:

1. Evidence of physical dependence on alcohol or benzodiazepines based on tolerance and withdrawal upon cessation of use of alcohol or benzodiazepines reported in the Mini-International Neuropsychiatric Interview (MINI) as well as clinical interviews by medical staff during H&P.
2. Seeking treatment for alcohol or substance use
3. Have a current physical or mental illness judged by the study team to negatively impact participant safety or scientific integrity
4. Active hepatic disease or abnormal liver function tests
5. Current major depressive disorder or suicidality
6. Are currently pregnant, planning to become pregnant in the next three months or are currently breastfeeding. People of childbearing potential will be asked to ensure, and/or the partner use effective forms of contraception for the duration of the study and excluded if unable.
7. Are currently enrolled in another clinical trial or have received any drug as part of a research study within 30 days of study participation.
8. Contraindications or allergies to study medications
9. Evidence of recent illicit substance use (i.e., positive urinalysis) at screening for drugs other than cannabis
10. Seizure disorder or traumatic brain injury (TBI)
11. Taking medications known to interact with study medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Demand Intensity - Consumption of Blinded Drug at Unconstrained Price as Measured by a Demand Task | Upon completion of experimental session (~8 hours post drug administration)
  Consumption of blinded drug at unconstrained price as measured by a demand task. Minimum value is 0, maximum value is not constrained. Higher scores indicate more drug consumption at unconstrained price (a worse outcome).
Breakpoint - Maximum price paid for blinded drug as measured by a demand task | Upon completion of experimental session (~8 hours post drug administration)
  Maximum price paid for blinded drug as measured by a demand task. Minimum value is 0, maximum value is not constrained. Higher scores indicate higher price paid (a worse outcome).
Cold Pressor Pain - Seconds to withdraw hand from cold pressor | Baseline and 1, 2, 4, and 6 hours post drug administration
  Seconds to withdraw hand from cold pressor laboratory pain task, where longer time periods reflect higher tolerance to pain.
Cognitive Performance assessed by Digit Symbol Substitution Test (DSST) | Baseline and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, and 8 hours post drug administration.
  Within-subject comparison of study conditions on the Digit Symbol Substitution Test (DSST), a measure of cognitive performance that is sensitive to drug effects, wherein lower percent scores reflect worse performance and suggest greater drug-related impairment.

SECONDARY OUTCOMES:
Drug Liking assessed by Visual Analog Scale of Drug Liking | Upon completion of experimental session (~9 hours post drug administration)
  Ratings on a visual analog scale of drug liking. Minimum value is 0 and maximum value is 100. Higher scores indicate greater drug liking (a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Justin Stricklahd, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Baltimore, Maryland, United States